CLINICAL TRIAL: NCT06786520
Title: A Phase 1 Single Arm, Repeat Dose Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Switching to Cabotegravir Ultra Long-acting From Cabotegravir Long-acting in Healthy Adult Volunteers
Brief Title: A Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of Cabotegravir Ultra Long-acting (CAB ULA) Following Switch From Cabotegravir Long-acting (CAB LA) in Healthy Adults
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 223369
Record Dates: First submitted 2025-01-15; First posted 2025-01-22 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: HIV Infections
Keywords: Cabotegravir (CAB); Ultra Long Acting (ULA); Long Acting (LA); Pharmacokinetics; Safety; Tolerability; Healthy Adult
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CAB Group (Experimental): Participants will receive the CAB LA Q2M regimen up to Month 9 then will receive the CAB ULA Q4M regimen up to Month 23.
  Interventions: Drug: CAB LA; Drug: CAB ULA

INTERVENTIONS:
Drug: CAB LA — CAB LA injection will be administered
Drug: CAB ULA — CAB ULA injection will be administered

SUMMARY:
This study will assess the pharmacokinetics (PK), safety, and tolerability of CAB ULA administered every 4 months (Q4M) following administration of CAB LA every 2 months (Q2M), in healthy adult volunteers.

DETAILED DESCRIPTION:
The participants in the study will receive CAB LA in the CAB LA phase and CAB ULA in the CAB ULA phase.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants greater than or equal to (>=) 18 years old, weighing at least 35 kg.
* Participants who are overtly healthy as determined by medical evaluation.
* Assigned male sex at birth or assigned female sex at birth. Participants assigned female sex at birth are eligible to participate if they are of non-childbearing potential, or if they are of childbearing potential and are not pregnant (confirmed by test), not breastfeeding, and are using a highly effective contraceptive method.
* Capable of giving written informed consent.

Healthcare staff will be eligible for inclusion in this study if:

* They are site employees responsible for administrative or clinical aspects of offering and administering CAB under the protocol at the site.
* Has the required qualifications according to their role and delegated the appropriate responsibilities by site Principal investigator (PI).
* Be able to understand and comply with protocol requirements, instructions, and restrictions.

Exclusion Criteria:

* Presence or history of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, haematological, neurological, or psychiatric disorders capable of significantly altering drug pharmacokinetics, interfering with the participant's ability to comply with the dosing schedule and/or protocol evaluations, or compromising participant safety.
* Current or anticipated need for chronic anti-coagulants.
* Any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.
* History of ongoing or clinically relevant seizure disorder within the previous 2 years.
* Participants who pose a significant suicidality risk.
* History or presence of sensitivity to any of the study medications, study procedure-related medications, their components or drugs of their class, or an allergy that contraindicates participation.
* Participant has an implant/enhancement (including fillers) at the area of proposed injection; or tattoo or other dermatological condition overlying any area which may significantly interfere with interpretation of injection site reactions.
* Inflammatory skin conditions that compromise the safety of injections.
* Any acute laboratory abnormality that should preclude participation or exclusionary laboratory value.
* Human immunodeficiency virus (HIV-1 or HIV-2) infection.
* Reactive or positive HIV test.
* Signs and symptoms suggestive of acute HIV infection- that is not ruled out with non-reactive results using appropriate HIV tests.
* Presence of hepatitis B surface antigen (HBsAg) at screening or within 3 months prior to first dose of study intervention.
* Positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study intervention.
* Positive hepatitis C RNA test result at screening or within 3 months prior to first dose of study intervention.
* One or more exclusionary values for a screening ECG.
* Participants receiving any protocol-prohibited medication.
* Use of CAB LA for PrEP within 1 year.
* Concurrent participation in another clinical study in which an investigational product was received within 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Participation in the study would result in loss of blood or blood products in excess of 500 mL within 56 days.
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* Positive pre-study drug/alcohol screen.
* History of or on-going high-risk behaviours that put the participant at increased risk for HIV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2025-01-17 (Actual); Primary Completion 2027-03-09 (Estimated); Study Completion 2027-11-08 (Estimated)

PRIMARY OUTCOMES:
Plasma concentration of CAB at the end of the CAB LA phase compared to plasma concentration of CAB at the end of the CAB ULA phase | At Month 23 compared to Month 9

SECONDARY OUTCOMES:
Plasma concentration of CAB at each assessment timepoint following CAB ULA injections | Up to Month 23
Number of participants with adverse events (AEs) (including Injection Site Reactions [ISRs]) as per severity | Up to Month 32
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. Severity is graded according to the Division of Acquired Immunodeficiency Syndrome (DAIDS) grading criteria, where Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = potentially life-threatening.
Number of participants with laboratory abnormalities | Up to Month 32
Number of participants with changes in laboratory parameters over time | Up to Month 32
Number of participants with ISRs by grade | Up to Month 32
  Severity of ISRs is graded according to the DAIDS grading criteria, where Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = potentially life-threatening
Duration (Days) of ISRs by grade | Up to Month 32
  Severity of ISRs is graded according to the DAIDS grading criteria, where Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = potentially life-threatening.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Oak Brook, Illinois

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.viiv-studyregister.com/documents/About_ViiV_Patient_Level_Data_Sharing_Final_25Sep2023.pdf